CLINICAL TRIAL: NCT06145646
Title: Influence of Intramuscular Temperature on the Textural Characteristics of the B-mode Ultrasound Image.
Brief Title: Intramuscular Temperature on the Echo-textural Characteristics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEEI23_453
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-02

CONDITIONS: Healthy Subjects
Keywords: muscle; temperature; texture; ultrasound; echo intensity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Muscle temperature (Experimental): Heating the vastus lateralis of the right quadriceps using microwaves
  Interventions: Device: Muscle warm-up

INTERVENTIONS:
Device: Muscle warm-up — Passive heating of the vastus lateralis of the right quadriceps will be performed using a microwave device. The device will be set at a power of 150 W and a distance of 10-15 cm from the skin surface for 20 minutes with the purpose of increasing local muscle temperature to 40 ºC.

SUMMARY:
Echointensity and echotexture have been used as a physiological marker for changes in skeletal muscle quality and structure caused by physical training, low activity, ageing and some neuromuscular disorders. However, there are some influencing factors on muscle echo-intensity and echotexture, such as temperature, which may not be taken into account when performing an ultrasound assessment and may alter the results.

This study aims to investigate the effects of muscle temperature on echointensity and other 2nd order echotextures variables such as homogeneity, contrast, correlation and entropy of muscle tissue, in order to gain a better understanding of this correlation and minimise its influence, which would allow greater precision in the use of muscle ultrasound as a diagnostic tool.

The methodology of this study includes firstly the acquisition of ultrasound images of the vastus lateralis muscle. This acquisition will be performed during the continuous recording of muscle temperature, carried out during a passive cooling process after 20 min of heating using microwave equipment. In addition, to standardise the results, a correction factor will be calculated to compensate for the influence of subcutaneous adipose tissue thickness on echogenicity and echotexture.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance of participation in the study.
* Healthy subjects.
* Subjects between the ages of 18 and 65.

Exclusion Criteria:

* Have known neurological, cardiovascular, metabolic or orthopedic conditions that prevent them from participating in the study.
* Present metal implants in the heating area.
* Wear a pacemaker.
* Perform physical activity during the 48 hours prior to data collection.
* Contraindications of dry needling such as: Belonephobia, history of abnormal reaction to the puncture or injection, anticoagulant treatment or thrombocytopenia, lymphedema over the area of intervention, severely compromised immune system, vascular diseases, diabetes mellitus, pregnancy, epilepsy, allergy to metals or that the intervention area has wounds, scars, tattoos, or stains.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Muscle echointensity (0-255 a.u.). | During intervention
  Muscle echointensity is calculated by the mean gray level value of the muscle Range of Interest (ROI). (0-255 a.u.)
Muscle echovariance (0-255 a.u.). | During intervention
  The echovariance is determined by the relationship between the standard deviation and the average pixel intensity obtained from the histogram of the muscle ROI. (0-255 a.u.)
Muscle energy or second angular momentum. | During intervention
  It is a second order parameter (GLCM) that measures textural uniformity of the muscle ROI
Muscle homogeneity. | During intervention
  It is a second-order parameter (GLCM) that measures the uniformity of the muscle ROI composition.
Contrast. | During intervention
  It is a second-order parameter (GLCM) that measures local variations in gray levels of the muscle ROI.
Textural Correlation. | During intervention
  It is a second-order parameter (GLCM) that expresses linear gray-level dependencies of the muscle ROI.
Entropy. | During intervention
  It is a second-order parameter (GLCM) to measure muscle ROI disorder.
Echointensity correction factor for adipose thickness | Pre-intervention
  The measurement of subcutaneous adipose thickness will be carried out through the average of the distance from the skin to the aponeurosis coinciding with the superficial interface of the muscle and with different pressures of the probe on the skin. This measure will be used to develop a correction factor that allows compensating the influence of this variable on echogenicity and echotexture, standardizing the results.
Muscle temperature (ºC). | Pre-intervention and during intervention
  Measurement of intramuscular temperature of the right vastus lateralis of the quadriceps (ºC)

SECONDARY OUTCOMES:
Age (years) | Pre-intervention
  Subject's age (years)
Sex (female or male) | Pre-intervention
  Subject's sex (female or male)
Dominance | Pre-intervention
  Dominant leg (right-left)
Body mass index | Pre-intervention
  It is a measure of body fat based on height and weight that applies to adult men and women

CONTACTS AND LOCATIONS:
Locations (1):
- Sergio Montero Navarro, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
Access to identified personal information will be restricted to the principal investigator of the study/collaborators, the Research Ethics Committee and authorized personnel, when necessary to verify the data and procedures of the study, but always maintaining their confidentiality in accordance to current legislation.
  The personal data of the participants, obtained during their participation in the project, will be kept for the time necessary for the development of this research, which is estimated to be 6 months, and will subsequently be destroyed, and cannot be kept without having previously been anonymized.

REFERENCES:
- [Background] Akima H, Yoshiko A, Tomita A, Ando R, Saito A, Ogawa M, Kondo S, Tanaka NI. Relationship between quadriceps echo intensity and functional and morphological characteristics in older men and women. Arch Gerontol Geriatr. 2017 May-Jun;70:105-111. doi: 10.1016/j.archger.2017.01.014. Epub 2017 Jan 20. PMID 28126635
- [Background] Young HJ, Jenkins NT, Zhao Q, Mccully KK. Measurement of intramuscular fat by muscle echo intensity. Muscle Nerve. 2015 Dec;52(6):963-71. doi: 10.1002/mus.24656. Epub 2015 Sep 7. PMID 25787260
- [Background] Pillen S, Tak RO, Zwarts MJ, Lammens MM, Verrijp KN, Arts IM, van der Laak JA, Hoogerbrugge PM, van Engelen BG, Verrips A. Skeletal muscle ultrasound: correlation between fibrous tissue and echo intensity. Ultrasound Med Biol. 2009 Mar;35(3):443-6. doi: 10.1016/j.ultrasmedbio.2008.09.016. Epub 2008 Dec 10. PMID 19081667
- [Background] Teixeira CA, Alvarenga AV, Cortela G, von Kruger MA, Pereira WC. Feasibility of non-invasive temperature estimation by the assessment of the average gray-level content of B-mode images. Ultrasonics. 2014 Aug;54(6):1692-702. doi: 10.1016/j.ultras.2014.02.021. Epub 2014 Mar 1. PMID 24630851
- [Background] Pinto MD, Silveira Pinto R, Nosaka K, Blazevich AJ. Do Intramuscular Temperature and Fascicle Angle Affect Ultrasound Echo Intensity Values? Med Sci Sports Exerc. 2023 Apr 1;55(4):740-750. doi: 10.1249/MSS.0000000000003082. Epub 2022 Nov 8. PMID 36355345
- [Background] Kenny GP, Reardon FD, Zaleski W, Reardon ML, Haman F, Ducharme MB. Muscle temperature transients before, during, and after exercise measured using an intramuscular multisensor probe. J Appl Physiol (1985). 2003 Jun;94(6):2350-7. doi: 10.1152/japplphysiol.01107.2002. Epub 2003 Feb 21. PMID 12598487
- See also: Description The University CEU-Cardenal Herrera is th first private university in the Valencian Community. It belongs to the Foundation San Pablo - CEU and is the leading educational organization in Spain with three Universities all over Spain — http://www.uchceu.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-11-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT06145646/Prot_SAP_ICF_000.pdf